CLINICAL TRIAL: NCT02993094
Title: Ixazomib (MLN9708) in Combination With Carboplatin in Pretreated Women With Advanced Triple Negative Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to slow recruitment, the study had to be terminated prematurely.
Sponsor: Arbeitsgemeinschaft medikamentoese Tumortherapie (Other)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGMT_MBC-10 (X16087); 2016-001421-13 (EudraCT Number)
Record Dates: First submitted 2016-12-04; First posted 2016-12-15 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Triple-Negative Breast Cancer
Keywords: breast cancer; advanced triple negative; ixazomib; carboplatin; CARIXA; Study Group of Medical Tumor Therapy (AGMT)
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — ixazomib; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ixazomib/Carboplatin (Experimental): Accelerated dose-escalation phase with a single-patient cohort per dose level until defined DLT is observed during cycle 1, or until dose level 4 is reached. At this dose level the cohort is expanded to three patients and dose escalation reverts to a conventional 3+3 escalation design.
  Intervention (experimental): Ixazomib; po; 3mg escalated to 4mg; day 1, 8, 15 Intervention (backbone): AUC 1.5 escalated to AUC 2.5; day 1, 8, 15
  Interventions: Drug: Ixazomib; Drug: Carboplatin

INTERVENTIONS:
Drug: Ixazomib — Cycles will be repeated every four weeks. All subjects will continue on study drug until disease progression, unacceptable toxicity or treatment discontinuation for any other reason.
  Other Names: MLN9708
Drug: Carboplatin — Cycles will be repeated every four weeks. Cycles will be repeated every four weeks. All subjects will continue on study drug until disease progression, unacceptable toxicity or treatment discontinuation for any other reason.

SUMMARY:
This is an open-label phase I/II study for patients with advanced (locally advanced inoperable or metastatic) triple-negative breast cancer progressing after first-line therapy receiving ixazomib on days 1, 8, and 15 in combination with carboplatin on days 1, 8, and 15. Cycles will be repeated every four weeks.

DETAILED DESCRIPTION:
The phase I part of this study uses an alternate dose escalation accelerated titration design. In the accelerated dose-escalation phase a single-patient cohort per dose level will be enrolled, until one dose limiting toxicity (DLT) or 2 moderate toxicities are observed during cycle 1, or until dose level 4 is reached. At this dose level the cohort is expanded to three patients and dose escalation reverts to a conventional 3+3 escalation design.

DLTs are defined as inability to deliver the drug combination of ixazomib and carboplatin due to drug related toxicity.

The maximum-administered dose (MAD) is defined as the dose at which DLT occur in at least two of six patients treated at that dose level. The dose just below the MAD is considered the maximum-tolerated dose (MTD), providing that DLT is observed in fewer than two of six treated patients (or fewer than one third if more than six patients will be treated) at that dose level. Determination of MAD and MTD is based on DLT observed during the first treatment cycle.

Phase II:

After establishing MTD in phase I, accrual continues to evaluate the efficacy and safety of the combination. A total of 41 patients will be included (patients enrolled in the phase I part within the conventional dose escalation phase at the dose level considered as the MTD may be included).

All subjects will continue on study drugs until disease progression, unacceptable toxicity or treatment discontinuation for any other reason.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or locally advanced (without curative loco-regional treatment options with curative intention) adenocarcinoma of the breast, histologically confirmed
* Triple-negative subtype defined as the absence of staining for estrogen receptor (IHC <1%), progesterone receptor (IHC <1%) and HER2/neu (IHC 1+ or ISH ratio of < 2.0 between Her2 gene copy number and centromere of chromosome 17 or a copy number of 4 or less)
* Signed informed consent prior to any study-specific procedure, with the understanding that consent may be withdrawn at any time without prejudice to future medical care
* Female patients, age ≥ 18 years
* At least one prior line of chemotherapy for metastatic or locally advanced disease or disease progression within 12 months of completion of adjuvant chemotherapy
* Documented disease progression
* At least one measurable lesion according to RECIST 1.1 criteria
* Life expectancy of at least 12 weeks
* Performance status ECOG 0-2
* Adequate left ventricular ejection fraction at baseline, defined as LVEF ≥ 50% by either echocardiogram or MUGA
* Peripheral neuropathy NCI CTCAE grade ≤ 1 or grade 2 if no pain on clinical examination
* Adequate hematological, liver and renal function:

Exclusion Criteria:

* Pregnant or lactating women
* Serious medical or psychiatric disorders that would interfere with the patient's safety or informed consent
* Clinically significant cardiovascular disease, requiring medication during the study and which might interfere with regularity of the study treatment, or not controlled by medication.
* Radiation of the target lesion within the last 4 weeks prior to randomization
* Prior radiation to ≥ 30% of bone marrow
* Active bacterial, viral or fungal infection
* Known HCV infection
* Patients with clinically apparent brain metastases or evidence of a spinal cord compression
* Major surgery within 14 days before enrollment
* Systemic treatment, within 14 days before the first dose of ixazomib, with strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort.
* Participation in other clinical trials, including those with other investigational agents not included in this trial, within 30 days of the start of this trial and throughout the duration of this trial
* Patients that have previously been treated with ixazomib, or participated in a study with ixazomib whether treated with ixazomib or not
* History of other malignancy; patients who have been disease-free for 5 years or patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible
* Prior treatment with a platinum derivative (except in (neo-)adjuvant setting if breast cancer recurrence did not occur within 12 months after (neo-)adjuvant chemotherapy completion) and/or with a proteasome inhibitor
* Known hypersensitivity to the study drugs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-11-21 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | From treatment start until MTD (12 months --> start Phase II Q3 2017)
  Determination of maximum tolerated dose (MTD) and dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Safety profile based on adverse events evaluation | During study treatment + 28 day after last study drug (approximately 3 years)
  Incidence, type, severity and consequences (e.g. study discontinuation) of an adverse event
Overall response rate | During study treatment every 8 weeks until progression + end of study treatment (approximately 3 years)
Clinical benefit rate | During study treatment every 8 weeks until progression + end of study treatment (approximately 3 years)
  Complete remission, partial remission or stable disease for at least 24 weeks
Progression-free survival (PFS) | During study treatment every 8 weeks until progression + end of study treatment (approximately 3 years)
Quality of Life of MBC patients | Baseline + every 8 weeks until progression + at end of study treatment (approximately 3 years)
  EORTC quality of life questionnaire (QLQ-C30 and QLQ-BR23)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Greil, MD, Study Director — PMU Salzburg: Universitätsklinik für Innere Medizin III
Locations (12):
- Austria (12):
  - Universitätsklinik für Innere Medizin Graz, Graz, Styria
  - Universitätsklinik für Frauenheilkunde Innsbruck, Innsbruck, Tyrol
  - Klinikum Kreuzschwestern Wels GmbH, Wels, Upper Austria
  - Landeskrankenhaus Feldkirch, Innere Med. II, Interne E, Feldkirch, Vorarlberg
  - UK Graz: Universitätsklinik für Frauenheilkunde und Geburtshilfe, Klinische Abteilung für Gynäkologie, Graz
  - LKH Hochsteiermark: Department für Hämato-Onkologie, Leoben
  - BHS Linz: Interne I: Internistische Onkologie, Hämatologie und Gastroenterologie, Linz
  - KUK Linz: Klinik für Interne 3 - Schwerpunkt Hämatologie und Onkologie, Linz
  - PMU Salzburg: Universitätsklinik für Innere Medizin III, Salzburg
  - Landeskrankenhaus Steyr, Innere Medizin II Onkologie, Steyr
  - AKH Wien Universitätsklinik für Frauenheilkunde: Klin. Abt. f. Allg. Gynäkologie und gynäkologische Onkologie, Vienna
  - LK Wiener Neustadt: Innere Medizin, Hämatologie und internistische Onkologie, Wiener Neustadt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rinnerthaler G, Gampenrieder SP, Petzer A, Burgstaller S, Fuchs D, Rossmann D, Balic M, Egle D, Rumpold H, Singer CF, Bartsch R, Petru E, Melchardt T, Ulmer H, Mlineritsch B, Greil R. Ixazomib in combination with carboplatin in pretreated women with advanced triple-negative breast cancer, a phase I/II trial of the AGMT (AGMT MBC-10 trial). BMC Cancer. 2018 Nov 6;18(1):1074. doi: 10.1186/s12885-018-4979-0. PMID 30400780